CLINICAL TRIAL: NCT07239258
Title: The Effects of Mir Shakeel Teleintegrated Therapy Plan and Conventional Physical Therapy on Pain, Range of Motion, Gait, Functional Outcomes and Quality of Life in Patients Undergoing Total Knee Arthroplasty
Brief Title: The Effects of Mir Shakeel Teleintegrated Therapy Plan on Pain, Range of Motion, Gait, Functional Outcomes and Quality of Life in Patients Undergoing Total Knee Arthroplasty
Acronym: RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mir Shakeel Ahmad (Other)
Responsible Party: Sponsor-Investigator, Mir Shakeel Ahmad, Principal Investigator, Lincoln University College
Organization: Lincoln University College (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHDMSTITPLUCGTTH24
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Total Knee Anthroplasty; Total Knee Arthroplasty Recovery
Keywords: pain; range of motion; gait; functional outcomes; quality of life; conventional physical therapy; total knee arthroplasty
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSTITP Group (Experimental): The patients of this group will be treated by the Physical Therapist in person as well as at Telerehabilitation mode as and when convenient for the patients. The treatment which shall be provided is a personalized exercise based treatment protocol already tested through a pilot testing on 80 patients in the same setting. This protocol is set under the supervision of an expert Orthopedic Surgeon from Ghurki Trust and Teaching Hospital. The protocol is composed of a weekly based exercise plan for patients who have underwent Total Knee Arthroplasty. The frequency and duration of each exercise is set owing to the age, severity and duration of surgery.
  Interventions: Other: Mir Shakeel Teleintegrated Therapy plan
- Conventional Physical Therapy (Active Comparator): The patients of this group will receive conventional physical therapy in which patients will have all sessions in person and within the premises of hospital/clinic. All the exercises and protocol provided to patients of experimental group will be practiced by patients of group B but no shift of exercise mode to Telerehabilitation will be made in order to rule out the effects of telerehabilitation if any.
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Mir Shakeel Teleintegrated Therapy plan — This intervention plan encompasses a weekly based exercise plan initated right from the Indoor patient department post surgery till week 23. It begins from within 24 hours of surgery and extends till 12 weeks post surgery. This includes sets of exercises in which the plan of week 1 includes patient education, bed mobility, transfers, ankle pumps, heel slides, straight reg raises, supine hip abduction and adduction, quads sets and seated knee flexion. Week 2 -4 include cryotherapy, ankle pumps, quad sets, heel slides, mini squats, standing heel raises, seated knee flexion and extension, marching in place and step ups. Week 4-6 include step ups, tandem walking, 3-d straight leg raises, sit to stand, single leg balance, mini squats, lunges, standing heel raises, marching with walker and toe raises while standing. Week 6-12 include single leg balance, gait training, single leg stand with trunk rotation, basu ball training, sideway walk and squats. This is encompassed by TR as &when needed.
  Arms: MSTITP Group
Other: Conventional Physical Therapy — The control group shall receive the same exercise plan in in - person treatment sessions 2-3 times per week. The set of exercises and frequency incorporated match with the one being provided to patients in group CPT.
  Arms: Conventional Physical Therapy

SUMMARY:
The objective of this clinical trial is to determine the effects of a newly formed treatment protocol implemented as telerehabilitation and compare it with conventional physical therapy in patient recovery after Total Knee Arthroplasty.

The main questions this study aims to answer are:

Does telerehabilitation improve pain, range of motion, and gait as effectively as conventional physical therapy?

Does telerehabilitation enhance exercise adherence, reduce kinesiophobia, and improve quality of life and patient satisfaction?

Can a hybrid rehabilitation protocol combining both approaches optimize clinical and functional outcomes?

Researcher will compare telerehabilitation-based physical therapy with traditional in-person therapy to see which method provides superior results in post-TKA recovery.

Participants Will:

Be adults aged 50-65 years who have undergone primary total knee arthroplasty

Receive either conventional physical therapy or a telerehabilitation-based exercise plan for a defined intervention period

Attend scheduled follow-up assessments to measure pain, range of motion, gait, functional performance, and satisfaction

Complete validated questionnaires on quality of life, kinesiophobia, and exercise adherence

Study Significance

Osteoarthritis is a growing health concern in Pakistan, with prevalence rising from 2.85 million in 1990 to 8.49 million in 2021. The increasing number of TKA procedures has created a demand for accessible, cost-effective, and evidence-based rehabilitation models. Telerehabilitation offers an innovative solution by extending professional care to patients' homes, enhancing accessibility, and ensuring continuity of therapy.

This study will provide locally relevant evidence and may lead to the development of a standardized rehabilitation protocol for Pakistani patients - improving recovery outcomes, reducing healthcare burden, and enhancing post-surgical quality of life

Ultimately, this research seeks to strengthen evidence-based rehabilitation in Pakistan, reduce the post-surgical burden of disability, and enhance the quality of life for individuals recovering from knee arthroplasty.

This RCT is based on a comparison of 2 groups. One will receive the MSTITP and other group will receive in person conventional physical therapy plan. This is based on 2 arm testing and the hypothesis is that the MSTITP is more effective in improving patient related outcomes in patients undergoing Total Knee Arthroplasty.

Participants in group A will perform a specific set of exercises ( details can be provided as and when asked) in a mode as convenient for the patients. The effect of Telerehabilitation will also be evaluated.

Participants in Group B will receive Conventional Physical Therapt as documented in in person sessions and will be followed for the same duration as of Patients in Group A.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have underwent a primary unilateral total knee arthroplasty due to osteoarthritis
* Able to participate in a rehabilitation program, either telerehabilitation or in-person, and demonstrate sufficient mobility with or without assistive devices (e.g., crutches, walker) as deemed appropriate for post-TKA therapy.
* Participants must have reliable access to a smartphone, tablet, or computer with internet connectivity and the ability to engage in video calls.
* Willing and able to provide informed consent, and to comply with all study protocols, including scheduled therapy sessions and follow-up assessments.

Exclusion Criteria:

* Presence of significant comorbidities or complications that could interfere with safe participation in rehabilitation, such as severe cardiovascular disease, or conditions causing significant immobility (e.g., severe osteoarthritis in other joints or Rheumatoid Arthritis.
* Previous knee replacement or other significant knee surgeries on the same knee, as this may impact the standardization of rehabilitation outcomes.
* Currently enrolled in another physical therapy or rehabilitation trial, or engaging in additional rehabilitation outside the study protocol.
* Cognitive impairment or severe visual or hearing impairments that would prevent them from following therapy instructions or engaging with telerehabilitation technology.
* Any other conditions or factors that, in the opinion of the investigators, could hinder compliance with the study procedures or put the participant at undue risk.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Both males and females will be allwed to particpate
Enrollment: 120 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | WEEK 1- WEEK 12
  Range of motion shall be measured through Goniometry
Pain of patient as assessed by Numerical Pain Rating Scale | Week 1 - Week 12
  The scale is composed of a scoring of 1 to 10 where 1 shows minimal pain and 10 shows maximal.
Quality of Life as assessed by Short Form Health Survey -36 | WEEK 1-WEEK 12
  SF 36 evaluates patient functions in 8 domains including physical functions, role limitations, body pain, health perceptions, vitality, social functions, role limitations and mental health. Higher schores reflect more functional impairements and lesser scores show less impairements. Each item is evaluated on a scale of 0-100.
Functional outcomes as assessed by Western Ontario and McMaster Universities Osteoarthritis Index | Week 1- Week 12
  The WOMAC is composed of 24 questions and scores from 0 to 96 where 0 reflects best health status
Gait as assessed through Jack's Observatory Gait Analysis | WEEK 1 - WEEK 12
  Gait analysis shall be done through Jacks' OGA

SECONDARY OUTCOMES:
Patient Satisfaction as assessed through Patient Satisfaction Questionnaire | WEEK 1- WEEK 12
  Patient Satisfaction shall be evaluated through PSQ-18 and it contains 18 items. Each item is scored from 1 to 5 and maximum score is 90 with 90 reflecting the best satisfaction levels of patients.
Exercise Adherence as assessed through Exercise Adherence Rating Scale | Week 1 - week 12
  Exercise adherence rating scale will be used to measure exercise adherence and the score ranges from 0-24. Higher scores reflect better exercise adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mir Shakeel Ahmad, PhD Scholar, Principal Investigator — Ghurki Trust and Teaching Hospital
Locations (1):
- Ghurki Trust and Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided